CLINICAL TRIAL: NCT05511688
Title: National Cohort of Colorectal Cancers With Microsatellite Instability
Status: Active, not recruiting | Type: Observational
Sponsor: Federation Francophone de Cancerologie Digestive (Other)
Responsible Party: Sponsor
Other Study IDs: Colomin2 Cohort
Record Dates: First submitted 2022-03-24; First posted 2022-08-23 (Actual); Last update posted 2025-09-02 (Actual); Status verified 2025-08

CONDITIONS: Colorectal Cancer; Microsatellite Instability
MeSH Terms: conditions — Colorectal Neoplasms; Microsatellite Instability

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

SUMMARY:
The three main pathways of colorectal carcinogenesis are chromosomal instability, microsatellite instability (MSI) (15% of colorectal cancers =CRCs) and CpG island methylator phenotype (CIMP). MSI CRCs are associated with a better prognosis after curative surgery than CRCs without microsatellite instability (MSS). In contrast, MSI CRCs do not appear to benefit from adjuvant 5-FU chemotherapy, unlike patients with MSS CRCs. Nevertheless, the benefit of adjuvant chemotherapy with FOLFOX seems to be retained. The identification of prognostic markers in this subgroup of patients is therefore essential to decide on adjuvant chemotherapy, the efficacy of which is currently debated in MSI CRC.

To date, there are very few data concerning metastatic MSI CRC. Metastatic forms are rare (about 5% of metastatic CRCs), but are thought to be associated with chemoresistance and poor prognosis. Nevertheless, data are very sparse and there are no data regarding the use of modern chemotherapies and targeted therapies in metastatic MSI CRC. Thus, it is important to characterize the chemosensitivity of metastatic forms.

Clinical predictors of recurrence after curative CRC surgery are known but have only been studied in MSI CRC retrospectively. Similarly, many molecular and immunohistochemical factors, prognostic or predictive of response to adjuvant chemotherapy, have been recently identified in CRC (KRAS, BRAF, TP53, PI3KCA mutations, CIMP phenotype, SMAD4, immune response...). Most of these markers have been studied in all CRCs, but not specifically in the MSI CRC subgroup. All these prognostic and/or predictive biomarkers need to be better characterized in a large cohort of MSI CRCs.

DETAILED DESCRIPTION:
Colorectal cancers with microsatellite instability The 3 main pathways of colorectal carcinogenesis are chromosomal instability (75% of CRCs), microsatellite instability (15% of CRCs) and CpG island hypermethylation or CIMP (CpG island methylator phenotype) (25% of CRCs).

Microsatellite instability (MSI) or RER+ (replication errors) phenotype is related to an acquired or inherited inactivation of the MMR (mismatch repair) system of DNA mismatch repair. In MSI CRCs associated with Lynch syndrome or HNPCC (hereditary nonpolyposis colorectal cancer) (3% of CRCs), there is a germline mutation in one of the genes of the MMR system, essentially MLH1 or MSH2, more rarely MSH6 or PMS2. In sporadic MSI cancers, frequently observed in the elderly, the loss of function of the MMR system is linked to a biallelic hypermethylation of the CpG islands of the MLH1 gene promoter causing its inactivation. Molecular individualization of CRCs has allowed the identification of tumor subgroups, such as MSI CRCs, that are more homogeneous in terms of their progression pathway, but the impact in terms of prognosis and treatment sensitivity remains to be clarified.

Prognosis and chemosensitivity of colorectal cancers with microsatellite instability MSI CRCs are associated with a better prognosis after curative surgery than CRCs without microsatellite instability (MSS) . In contrast, retrospective analyses of randomized trials indicate that patients with MSI CRC do not appear to benefit from adjuvant 5-FU-based chemotherapy in contrast to patients with MSS CRC. Nevertheless, the benefit of adjuvant chemotherapy with FOLFOX seems to be retained . The identification of prognostic markers in this subgroup of patients is therefore essential to decide on adjuvant chemotherapy, the efficacy of which is currently debated in MSI CRC.

To date, there are very few data concerning metastatic MSI CRC. Metastatic forms are rare (about 5% of metastatic CRCs), but are thought to be associated with chemoresistance and poor prognosis . Nevertheless, data are very sparse and there are no data regarding the use of modern chemotherapies and targeted therapies in metastatic MSI CRC. Thus, it is important to characterize the chemosensitivity of metastatic forms in order to offer the best treatment to patients.

Recent data show significant efficacy of immune checkpoint inhibitors in MSI CRC, including anti-PD1. Indeed, these tumors present a high number of mutations generating immunogenic neo-antigens. Thus, escape from anti-tumor immunity is a major mechanism of progression of MSI CRCs .

Prognostic and predictive factors of response to chemotherapy in colorectal cancer with microsatellite instability The clinical predictive factors for recurrence after curative CRC surgery are known (lymph node involvement, T4 stage, VELIPI criteria (vascular emboli, perineural sheaths, and lymphatic emboli), poorly differentiated tumor, analysis of fewer than 12 nodes, tumor perforation, and overt bowel obstruction). These criteria have only been studied in MSI CRCs retrospectively. A large French retrospective study of MSI CRCs included 521 MSI CRCs. Four independent predictors of recurrence-free survival were identified, age (HR=1.02; 95%IC 1.00-1.04, p=0.014), initial bowel obstruction (HR=2.33; 95%CI 1.29-4.23, p=0.005), vascular emboli (HR=2.27; 95%IC 1.41-3.63, p<0.001), and stage T4 (HR=2.09; 95%IC 1.28-3.40, p=0.003). It should be noted that, unlike MSS CRCs, the prognostic impact of lymph node involvement appears to be small. This work is nevertheless limited by missing data (5-30%), biases related to retrospective analysis and the absence of exploitable molecular analyses (notably KRAS and BRAF mutation). These data can be validated prospectively from the COLOMIN 2 cohort.

In stage III MSI CRC, adjuvant chemotherapy with FOLFOX is recommended. On the other hand, in stage II MSI CRC, simple surveillance is recommended given the good prognosis . Nevertheless, in case of vascular emboli and/or T4 stage in MSI stage II CRC, the risk of recurrence becomes clinically significant (more than 20% at 2 years) and therefore raises the question of adjuvant treatment on a case-by-case basis. Indeed, in high-risk stage II MSI CRC, FOLFOX seems to provide a benefit in terms of recurrence-free survival compared with surgery alone . The COLOMIN 2 cohort will allow prospective confirmation of the chemosensitivity of these tumors to oxaliplatin.

Many molecular and immunohistochemical factors, prognostic or predictive of response to adjuvant chemotherapy, have been recently identified in CRC (KRAS, BRAF, TP53, PI3KCA mutations, CIMP phenotype, SMAD4, immune response...). These markers have been mostly studied in all CRCs, but not specifically in the subgroup of MSI CRCs. All these molecular and immunohistochemical factors need to be better characterized in a large cohort of MSI CRCs in order to determine their exact frequencies, their associations with each other, their prognostic and predictive values of response to chemotherapy. The constitution of a biological collection in COLOMIN 2 will allow the analysis of different biomarkers. For example, the BRAF mutation (V600E) is associated with a poor prognosis in CRC. Nevertheless, its prognostic impact remains debated in MSI CRC, whereas more than 50% of MSI CRC are BRAF mutated. COLOMIN 2 will assess the prognostic impact of BRAF mutation in MSI CRC.

ELIGIBILITY:
Inclusion Criteria:

* Patient with MSI colorectal cancer defined either by molecular biology (more than 30% of microsatellites tested unstable) or by immunohistochemistry (loss of expression of at least one MMR protein: MLH1, MSH2, MSH6, PMS2)
* Histologically proven colorectal cancer diagnosed on or after January 1 of the cohort start date
* Stage I, II, III (non-metastatic) or IV (metastatic)

Exclusion Criteria:

* Colorectal cancer MSS
* Contraindication due to psychological, social, or geographical reasons that may hinder patient follow-up
* Opposition of the patient to registration in the cohort
* Stage 0 (Tumor in situ, N0, M0)

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients with MSI colrectal cancers (stage I to IV)
Sampling Method: Non-Probability Sample
Enrollment: 637 (Actual)
Dates: Start 2017-03-22 (Actual); Primary Completion 2025-12 (Estimated); Study Completion 2025-12 (Estimated)

PRIMARY OUTCOMES:
Progression Free Survival for stage IV colorectal cancers | from date of diagnosis up to 36 months
  Identification of clinical, immunohistochemical and molecular prognostic factors
Time to recurrence for stage I , II or III colorectal cancers | from date of diagnosis up to 36 months
  Identification of clinical, immunohistochemical and molecular prognostic factors

CONTACTS AND LOCATIONS:
Overall Officials: David Tougeron, MD PHD, Principal Investigator — CHU POTIERS
Locations (14):
- France (14):
  - Chu Poitiers, Poitiers, VIENNE
  - CH, Abbeville
  - Chu - Hôpital Sud, Amiens
  - Chu - Hôpital Hôtel Dieu, Angers
  - CH, Angoulême
  - Ch - Hôpital Victor Dupouy, Argenteuil
  - Ch - Ght Unyon Auxerre, Auxerre
  - Ch - Hôpital Henri Duffaut, Avignon
  - Privé - Institut Du Cancer Avignon Provence, Avignon
  - Chu - Hôpital Jean Minjoz, Besançon
  - Privé- Centre Pierre Curie, Beuvry
  - Ch - Centre Hospitalier de Bézier, Béziers
  - Privé - Clinique Tivoli, Bordeaux
  - Privé - Polyclinique Bordeaux Nord, Bordeaux

IPD SHARING:
Plan to Share IPD: Undecided